CLINICAL TRIAL: NCT00388817
Title: Improving Medication Use in Patients With Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Indiana University School of Medicine (Other); Wishard Health Services (Other)
Organization: University of North Carolina, Chapel Hill (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01HL069399 (NIH)
Record Dates: First submitted 2006-10-08; First posted 2006-10-17 (Estimated); Last update posted 2006-10-17 (Estimated); Status verified 2006-10

CONDITIONS: Hypertension
Keywords: Hypertension; Blood pressure; Adherence; Compliance; Pharmacist; Pharmacy; Costs
MeSH Terms: conditions — Hypertension; Patient Compliance

INTERVENTIONS:
Behavioral: Pharmacist intervention

SUMMARY:
The purpose of this trial is to determine whether minority and low-income patients with high blood pressure take their medications better when they are helped by a pharmacist and provided with special medication packaging and information aimed at persons with low health literacy.

DETAILED DESCRIPTION:
Optimal use of medications in patients with hypertension prevents adverse outcomes. When their blood pressure is carefully controlled, patients with uncomplicated hypertension are spared primary events including myocardial infarction, stroke, cognitive impairment, and renal insufficiency. Patients who have already experienced complications are spared the suffering of subsequent events. Because hypertension is asymptomatic and antihypertensive drugs have adverse effects, patients often feel better when they are not taking their medication as opposed to when they carefully adhere to their physician's prescribed regimen. Therefore, innovative strategies are needed to educate patients and improve patient adherence to a complicated regimen often involving many drugs. Doing so can to reduce morbidity, mortality, and the costs of patient care. Minority patients often do not have access to the resources needed to assist them with their medications and as such they are especially vulnerable. Recent studies suggest that blood pressure control of patients with hypertension improves when pharmacists provide patients with education and monitoring. However, studies of clinical endpoints have not been conducted. This study aims to develop and test, in a randomized controlled trial, a multileveled pharmacy-based program to improve adherence in minority patients. This program incorporates patient education materials and medication packaging designed for patients with low-literacy. A study pharmacist accessed a computer database that is integrated into an electronic medical database called the Regenstrief Medical Record System (RMRS).

Patients from Wishard Health Services with uncomplicated or complicated hypertension were randomly assigned to a pharmacist intervention or usual care group. Patients in the intervention group received verbal education, written education materials, icon-based labeling of medication containers, and therapeutic monitoring. The pharmacist educated patients about their medications, identified barriers to appropriate drug use, coached patients to overcome drug use barriers, and coordinated drug use for these patients in conjunction with their primary care providers. Patients in the usual care (control) group did not receive pharmacist intervention.

To objectively measure medication compliance, Medication Event Monitor System (MEMS) lids (electronic monitors) were used for all antihypertensive medications. MEMS lids contain a computer chip that electronically imprints a time/date stamp each time an opening and closure occurs. Such data reveal the temporal pattern of medication adherence. Data concerning clinical endpoints, comorbidities, and healthcare costs were extracted from the RMRS. Other data included blood pressure measurements, health related quality of life, cognitive function, health literacy, and satisfaction with care.

Study participation for the patients in the intervention group concluded after 12 months of active intervention, which be followed by six months of post-intervention follow-up. Primary endpoints included medication adherence and systolic and diastolic blood pressures. Secondary outcomes included health-related quality of life, symptoms, patient satisfaction, and direct healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* plan to receive health care and prescriptions at study facility
* prescribed at least one blood pressure medication
* English-speaking
* access to a telephone
* no hearing impairments in the normal range of conversation

Exclusion Criteria:

* dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 492
Dates: Start 2002-01; Study Completion 2005-05

PRIMARY OUTCOMES:
Adherence to blood pressure medications
Blood pressure control

SECONDARY OUTCOMES:
Health-related quality of life
Exacerbation of symptoms
Patient satisfaction
Direct costs

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Murray, PharmD, MPH, Principal Investigator — UNC-Chapel Hill
Locations (1):
- School of Pharmacy, UNC-Chapel Hill, CB 7360, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Murray MD, Ritchey ME, Wu J, Tu W. Effect of a pharmacist on adverse drug events and medication errors in outpatients with cardiovascular disease. Arch Intern Med. 2009 Apr 27;169(8):757-63. doi: 10.1001/archinternmed.2009.59. PMID 19398687